CLINICAL TRIAL: NCT00023725
Title: A Randomized Phase I/II Study Of Preoperative Radiotherapy With/Without SUGEN 5416 (NSC # 696819; A TK Inhibitor Anti-Angiogenesis Compound) In The Management Of Low To Intermediate Grade Soft Tissue Sarcoma Of The Trunk or Extremity
Brief Title: Radiation Therapy With or Without SU5416 in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068854; RTOG-S-0120
Record Dates: First submitted 2001-09-13; First posted 2003-10-15 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2007-08

CONDITIONS: Sarcoma
Keywords: stage I adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Semaxinib; Radiotherapy

INTERVENTIONS:
Drug: semaxanib
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as SU5416 may stop the growth of cancer by stopping blood flow to the tumor. It is not yet known if radiation therapy is more effective with or without SU5416 in treating soft tissue sarcoma.

PURPOSE: Phase I/II trial to compare the effectiveness of radiation therapy with or without SU5416 in treating patients who have stage IB or stage IIA soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of SU5416 when combined with neoadjuvant radiotherapy in patients with stage IB or IIA soft tissue sarcoma.
* Determine the antiangiogenic effects of SU5416 in these patients.
* Determine any synergistic antiangiogenic effect of SU5416 with radiotherapy in these patients.
* Compare the disease-free survival, local recurrence, distant metastases, and overall survival rates in patients treated with neoadjuvant radiotherapy with or without SU5416.

OUTLINE: This is a phase I dose-escalation study of SU5416 followed by a phase II randomized study.

Phase I:

* Patients undergo radiotherapy once daily, 5 days a week, for 5 weeks. Patients also receive SU5416 IV over 1 hour twice weekly beginning on week 1 and continuing until 2 days before surgery.
* Cohorts of 3-6 patients receive escalating doses of SU5416 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Phase II:

* Once the MTD has been determined, additional patients are accrued and then randomized to receive either treatment as in phase I at the MTD vs preoperative radiotherapy alone.

All patients undergo surgical resection 70-80 days after beginning therapy. Patients with positive surgical margins receive additional radiotherapy daily for 8 days and SU5416 IV over 1 hour on days 2, 4, and 9.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 18 patients will be accrued for phase I of this study within 1 year. Approximately 28 patients will be accrued for phase II of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary or locally recurrent stage IB or IIA soft tissue sarcoma

  * Grade 1 or 2
  * Tumor greater than 5 cm in diameter
* Tumor located on upper extremities (including shoulder), lower extremities (including hip), or body wall
* No sarcoma of the head and neck or intra-abdominal or retroperitoneal sarcoma
* No desmoid tumor or dermatofibrosarcoma protuberans
* No metastatic disease
* No evidence of lung metastases

  * Maximum of 4 lung lesions no greater than 5 mm in diameter each on preoperative chest CT scan allowed OR
  * Lesion no greater than 1 cm allowed if stable for at least 1 year and fits criteria for granuloma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1

Life expectancy:

* At least 2 years

Hematopoietic:

* WBC at least 4,000/mm^3 OR
* Absolute neutrophil count at least 1,800/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 50 U/L
* PT and PTT less than 1.25 times normal (not on warfarin)

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* No congestive heart failure or myocardial infarction within the past 6 months
* No uncompensated coronary artery disease
* No severe peripheral vascular disease
* No peripheral vascular disease with diabetes mellitus
* No deep venous or arterial thrombosis within the past 3 months
* Fibrin split products less than 2 times normal
* Fibrinogen greater than 200 mg/dL

Pulmonary:

* No pulmonary embolism within the past 3 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindications to surgery
* No active uncontrolled bacterial, viral, or fungal infection
* No other prior or concurrent malignancy within the past 5 years except surgically treated carcinoma in situ of the cervix or squamous cell or basal cell skin cancer
* No other serious medical or psychiatric illness that would preclude informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for soft tissue sarcoma

Chemotherapy:

* No prior chemotherapy for soft tissue sarcoma

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for soft tissue sarcoma

Surgery:

* At least 2 weeks since prior minor surgery (e.g., port placement)
* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burton L. Eisenberg, MD, Study Chair — Fox Chase Cancer Center
Locations (226):
- United States (207):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscallosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mount Diablo Medical Center, Concord, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarian Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - Nebraska Health System, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fitzgerald Mercy Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon-Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (19):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan